CLINICAL TRIAL: NCT07091383
Title: The Effect of Instrument-Assisted Soft Tissue Mobilization on Pain, Skinfold Thickness, Shortness, and Functional Muscle Strength in Sedentary Individuals With Hamstring Tightness
Brief Title: The Effects of Instrument-Assisted Soft Tissue Mobilization in Sedentary Individuals With Hamstring Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus International University (Other)
Responsible Party: Principal Investigator, Mehmet Miçooğulları, Asst. Prof., Cyprus International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: -020-5432
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Hamstring Muscle Tightness; Muscle Strength; Pain Threshold
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The same physiotherapist will be administered all IASTM, functional IASTM, and static stretching interventions, while assessments will be conducted by another physiotherapist who will be blinded to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Static Stretching Group (Active Comparator): Participants will lie supine on a treatment table, with the non-test leg stabilized using a strap. Using a belt looped around the foot, the participant's ankle will be held in dorsiflexion, and passive hip flexion will be performed without knee flexion, stretching the hamstring to its maximal tension. The stretch will be held for 15 seconds and then relaxed. This cycle will be repeated 10 times per session.
  Interventions: Other: Exercise
- IASTM Group (Experimental): Participants will lie prone on the treatment table with their feet hanging off the edge. While the therapist holds the Graston tool in the right hand, passive knee flexion and extension movements will be performed with the left hand. After non-allergenic jelly is applied, the GT5 will be used to perform the sweep technique at a 30° angle along the hamstring for 10 repetitions, with one knee flexion during each sweep. The fan technique will then be applied in a similar manner, with knee flexion at each proximal movement. Subsequently, the GT4 will be used at a 60° angle for 10 repetitions of each sweep and fan technique, incorporating knee flexion with each proximal pass. Finally, the GT3 will be used to perform the brush technique at a 60° angle for 10 repetitions with knee flexion.
  Interventions: Other: Exercise
- Functional IASTM Group (Experimental): Participants will lie prone on the treatment table with their feet hanging off the edge. While the therapist holds the Graston tool in the right hand, passive knee flexion and extension movements will be performed with the left hand. After non-allergenic jelly is applied, the GT5 will be used to perform the sweep technique at a 30° angle along the hamstring for 10 repetitions, with one knee flexion during each sweep. The fan technique will then be applied in a similar manner, with knee flexion at each proximal movement. Subsequently, the GT4 will be used at a 60° angle for 10 repetitions of each sweep and fan technique, incorporating knee flexion with each proximal pass. Finally, the GT3 will be used to perform the brush technique at a 60° angle for 10 repetitions with knee flexion.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Static stretching
  Other Names: Stretching
  Arms: Static Stretching Group
Other: Exercise — Soft Tissue Mobilization
  Other Names: Soft Tissue mobilization
  Arms: IASTM Group
Other: Exercise — Functional soft tissue mobilization
  Other Names: Functional Soft Tissue Mobilization
  Arms: Functional IASTM Group

SUMMARY:
The aim of this study will be to investigate and compare the effects of static stretching exercise, Instrument Assisted Soft Tissue Mobilization (IASTM), and functional IASTM techniques on hamstring muscle shortness, pain threshold, skinfold thickness, and functional muscle strength in sedentary individuals. Fifty-one sedentary individuals between the ages of 18 and 45 who meet the inclusion criteria of Cyprus International University will be included in the study. The first group will receive static stretching exercises two days a week for four weeks; the second group will receive the IASTM technique two days a week for four weeks; and the third group will receive the functional IASTM technique, which will be applied with passive movements two days a week for four weeks. Hamstring shortness, pain threshold, skinfold thickness, and functional muscle strength will be evaluated before the treatment (BT), immediately after the treatment (AT1), two weeks after the treatment (AT2), and four weeks after the treatment (AT4).

ELIGIBILITY:
Inclusion Criteria:

* Sedentary individuals aged 18 to 45
* Who worked at a desk for extended periods
* Who exhibited hamstring muscle tightness of more than 10 degrees

Exclusion Criteria:

* Diagnosed orthopaedic or neurological disorder
* a history of lower limb surgery
* The presence of scoliosis
* Tightness in the gastrocnemius muscle
* Participants who did not consistently attend the intervention programme (i.e., those who missed two or more sessions out of the 12 sessions)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Hamstring Muscle Tightness | 4 weeks
  Hamstring tightness will be assessed using the PostureScreen Mobile application, a validated tool for photographic posture and joint angle analysis. Participants will lie supine on a treatment table with the non-test leg stabilized using a strap. The test leg will be positioned with both the hip and knee at 90° flexion, adjusted with a stool and pillow as needed. The anatomical landmarks-the greater trochanter, lateral femoral condyle, and lateral malleolus-will be marked on the test leg. While the participant wears minimal clothing, a lateral photograph will be taken from 1.5 metres using a tripod-mounted smartphone. Participants will be instructed to extend their knee as much as possible with their ankle dorsiflexed. The application will calculate the knee extension angle from the marked points, and the range of motion will be recorded in degrees. The test will be repeated if compensatory movements are observed.
Hamstring Skinfold Thickness | 4 weeks
  The site will be marked at the midpoint of the posterior thigh, halfway between the ischial tuberosity and the popliteal region. The skinfold will be grasped 1 cm from the marked point using the thumb and index finger, maintaining consistent pressure throughout the measurement. Skinfold thickness will be measured with a skinfold calliper (Holtain Ltd, Crymych, UK). The reading will be taken 3-4 seconds after applying the calliper and then recorded. At least two measurements will be taken with a one-minute interval between them. Results will be recorded in millimetres (mm).

SECONDARY OUTCOMES:
Pain Threshold | 4 weeks
  A pressure algometer will be used to assess the sensitivity of the area where pain is felt and to obtain a quantitative measure of pressure perception. In the assessment, a digital algometer (Algometer Commander, Jtech Medical, 801-478, USA) will be used. For the measurement, the participant will be positioned in the prone position. The motor point on the participant's hamstring muscle will be marked with a pen. The calibrated algometer, with a probe tip of 1 cm² diameter, will be placed perpendicularly on the marked point of the hamstring muscle. The physiotherapist will gradually apply pressure, and pressure will be increased until the participant perceives pain. Upon the participant's signal indicating pain, the pressure will be stopped and the probe will be removed. This test will be repeated three times, and the average value will be recorded.
Functional Muscle Strength | 4 weeks
  The "Five Times Sit-to-Stand Test" will be used to assess functional muscle strength. This test will evaluate the functional strength of the lower extremity, transitional movements, balance, and risk of falling. Participants will be asked to sit on a chair with a straight back and a seat height of 43-45 cm from the ground. They will be instructed to cross their arms over their chest, placing their hands on the opposite shoulders, and to stand up and sit down five times as quickly as possible without pausing. The test will begin with the participant standing, feet shoulder-width apart, and the trunk upright. Each complete sit-to-stand movement will be counted as one repetition. The time taken to complete five repetitions will be measured with a stopwatch and recorded in seconds. The stopwatch will be stopped when the participant stands up for the fifth time, and the result will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Cyprus International University, Mersin, Lefkosa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gallon D, Rodacki AL, Hernandez SG, Drabovski B, Outi T, Bittencourt LR, Gomes AR. The effects of stretching on the flexibility, muscle performance and functionality of institutionalized older women. Braz J Med Biol Res. 2011 Mar;44(3):229-35. doi: 10.1590/s0100-879x2011007500012. Epub 2011 Jan 26. PMID 21399855
- [Background] Kim J, Sung DJ, Lee J. Therapeutic effectiveness of instrument-assisted soft tissue mobilization for soft tissue injury: mechanisms and practical application. J Exerc Rehabil. 2017 Feb 28;13(1):12-22. doi: 10.12965/jer.1732824.412. eCollection 2017 Feb. PMID 28349028
- [Background] Markovic G. Acute effects of instrument assisted soft tissue mobilization vs. foam rolling on knee and hip range of motion in soccer players. J Bodyw Mov Ther. 2015 Oct;19(4):690-6. doi: 10.1016/j.jbmt.2015.04.010. Epub 2015 May 5. PMID 26592226
- [Background] Lee JH, Lee DK, Oh JS. The effect of Graston technique on the pain and range of motion in patients with chronic low back pain. J Phys Ther Sci. 2016 Jun;28(6):1852-5. doi: 10.1589/jpts.28.1852. Epub 2016 Jun 28. PMID 27390432
- [Background] Stutchfield BM, Coleman S. The relationships between hamstring flexibility, lumbar flexion, and low back pain in rowers. European Journal of Sport Science. 2006;6(4):255-260.
- [Background] Fatima G, Qamar MM, Hassan JU, Basharat A. Extended sitting can cause hamstring tightness. Saudi Journal of Sports Medicine. 2017;17(2):110-114.
- [Background] Afonso J, Rocha-Rodrigues S, Clemente FM, Aquino M, Nikolaidis PT, Sarmento H, Filter A, Olivares-Jabalera J, Ramirez-Campillo R. The Hamstrings: Anatomic and Physiologic Variations and Their Potential Relationships With Injury Risk. Front Physiol. 2021 Jul 7;12:694604. doi: 10.3389/fphys.2021.694604. eCollection 2021. PMID 34305648